CLINICAL TRIAL: NCT02051608
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multicenter, Efficacy and Safety Study of Gantenerumab in Patients With Mild Alzheimer's Disease; Part II: Open-Label Extension For Participating Patients
Brief Title: A Study of Gantenerumab in Participants With Mild Alzheimer Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WN28745; 2013-003390-95 (EudraCT Number)
Record Dates: First submitted 2014-01-30; First posted 2014-01-31 (Estimated); Results first posted 2022-06-16 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — gantenerumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1 (Double Blind treatment): Placebo (Placebo Comparator): Participants received matching placebo by subcutaneous (SC) injection every 4 weeks (Q4W) up to 100 weeks during Part 1 of the study.
  Interventions: Drug: Placebo
- Part 1 (Double Blind treatment): Gantenerumab (Experimental): Participants received 105 mg Gantenerumab by SC injection Q4W for 24 weeks and if eligible 225 mg SC injection Q4W from weeks 28-100 during Part 1 of the study.
  Interventions: Drug: Gantenerumab
- Part 2 (Open-Label Extension [OLE] treatment): Placebo switched to Gantenerumab Up to 1200 mg (Placebo Comparator): Participants who had received Placebo in Part 1, received Gantenerumab at doses up to 1200 mg by SC injection Q4W for up to 2 years. Additionally, participants were given the option to continue receiving open-label gantenerumab treatment for 3 years.
  Interventions: Drug: Placebo
- Part 2 (OLE treatment): Gantenerumab up to 1200 mg (Experimental): Participants who had received Gantenerumab in Part 1, received treatment at doses up to 1200 mg by SC injection Q4W for up to 2 years. Additionally, participants were given the option to continue receiving open-label gantenerumab treatment for 3 years.
  Interventions: Drug: Gantenerumab

INTERVENTIONS:
Drug: Placebo — Participants received Placebo SC injection Q4W.
  Arms: Part 1 (Double Blind treatment): Placebo; Part 2 (Open-Label Extension [OLE] treatment): Placebo switched to Gantenerumab Up to 1200 mg
Drug: Gantenerumab — Participants received Gantenerumab at 105 mg , 225 mg, or at doses up to 1200 mg SC injection Q4W.
  Arms: Part 1 (Double Blind treatment): Gantenerumab; Part 2 (OLE treatment): Gantenerumab up to 1200 mg

SUMMARY:
Part 1 is a multicenter, randomized, double-blind, placebo-controlled, parallel-group study will evaluate the efficacy and safety of gantenerumab in participants with mild Alzheimer disease. Participants will be randomized to receive either gantenerumab subcutaneously every 4 weeks or placebo subcutaneously every 4 weeks. Approved Alzheimer medication is allowed if on stable dose for 3 months prior to screening. Part 2 is an open-label extension (OLE).

A positron emission tomography (PET) imaging substudy will be conducted within the main study. Eligible participants who provide separate informed consent will undergo PET imaging scans using the radioligand florbetapir as a pharmacodynamic measure of changes in brain amyloid load over time.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of probable mild Alzheimer disease (AD) based on National Institute of Neurological and Communicative Disorders and Stroke/Alzheimer's Disease and Related Disorders Association (NINCDS/ADRDA) criteria or major NCD based whether or not receiving AD approved medication
* Cerebral spinal fluid (CSF) result consistent with the presence of amyloid pathology
* Availability of a person ('caregiver') who in the investigator's judgment has frequent and sufficient contact with the participant, and is able to provide accurate information regarding the participant's cognitive and functional abilities
* Fluency in the language of the tests used at the study site
* Willingness and ability to complete all aspects of the study
* Adequate visual and auditory acuity, in the investigator's judgment, sufficient to perform the neuropsychological testing (eye glasses and hearing aids are permitted)
* If currently receiving approved medications for AD, the dosing regimen must have been stable for 3 months prior to screening
* Agreement not to participate in other research studies for the duration of this trial and its associated substudies

PART 2 - All participants who have been randomized and are actively participating in the study are eligible for Part 2

Exclusion Criteria:

* Dementia or neurocognitive disorder (NCD) due to a condition other than AD, including, but not limited to, frontotemporal dementia, Parkinson disease, dementia with Lewy bodies, Huntington disease, or vascular dementia
* History or presence of clinically evident vascular disease potentially affecting the brain that in the opinion of the investigator has the potential to affect cognitive function
* History or presence of stroke within the past 2 years or documented history of transient ischemic attack within the last 12 months
* History or presence of systemic autoimmune disorders potentially causing progressive neurologic disease with associated cognitive deficits
* History of schizophrenia, schizoaffective disorder, or bipolar disorder
* Alcohol and/or substance use disorder (according to the DSM-5) within the past 2 years (nicotine use is allowed)
* History or presence of atrial fibrillation
* Within the last 2 years, unstable or clinically significant cardiovascular disease (e.g., myocardial infarction, angina pectoris, cardiac failure New York Heart Association Class II or higher)
* Uncontrolled hypertension
* Chronic kidney disease
* Impaired hepatic function

PET imaging substudy, in addition to above:

- Prior participation in other research study or clinical care within the last year such that the total radiation exposure would exceed the local or national annual limits

Part 2 Participants who have been discontinued from the study

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 389 (Actual)
Dates: Start 2014-03-27 (Actual); Primary Completion 2021-04-16 (Actual); Study Completion 2021-04-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (131):
- United States (30):
  - Banner Sun Health Research Insitute, Sun City, Arizona
  - Territory Neurology and Research Institute, Tucson, Arizona
  - ATP Clinical Research, Inc, Costa Mesa, California
  - Pacific Research Network - PRN, San Diego, California
  - California Neuroscience Research Medical Group, Inc, Sherman Oaks, California
  - Meridien Research, Brooksville, Florida
  - Brain Matters Research, Inc., Delray Beach, Florida
  - Neuropsychiatric Research; Center of Southwest Florida, Fort Myers, Florida
  - Miami Jewish Health Systems; Clinical Research, Miami, Florida
  - Accelerated Enrollment Solutions, Orlando, Florida
  - University of South Florida, Tampa, Florida
  - Alzheimer's Research and Treatment Center, Wellington, Florida
  - Indiana University, Indianapolis, Indiana
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana
  - Louisiana Research Associates, New Orleans, Louisiana
  - Western Michigan University Homer Stryker M.D. School of Medicine Center for Clinical Research, Kalamazoo, Michigan
  - Millennium Psychiatric Associates, LLC, St Louis, Missouri
  - Alzheimer's Research Corporation, Paterson, New Jersey
  - Ocean Rheumatology, Toms River, New Jersey
  - Nathan Kline Institute, Orangeburg, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - Alzheimer's Memory Center, Matthews, North Carolina
  - Richard H Weisler, MD, Raleigh, North Carolina
  - Central States Research, Tulsa, Oklahoma
  - Abington Neurological Associates, Abington, Pennsylvania
  - Northeastern Pennsylvania Memory, Plains, Pennsylvania
  - Rhode Island Mood & Memory Research Institute, East Providence, Rhode Island
  - Neurology Clinic PC, Cordova, Tennessee
  - Senior Adults Specialty Research, Austin, Texas
  - University of Utah, Center for Alzheimer's Care Imaging & Research, Salt Lake City, Utah
- Instituto Neurologia Bs As, Ciudad Autonoma Buenos Aires, Argentina
- Australia (4):
  - Royal Adelaide Hospital; Memory Trials Centre, Adelaide, South Australia
  - The Queen Elizabeth Hospital; Neurology, Woodville, South Australia
  - Heidelberg Repatriation Hospital; Medical and Cognitive Research Centre, Heidelberg West, Victoria
  - Australian Alzheimer's Research Foundation, Nedlands, Western Australia
- Belgium (2):
  - Cliniques Universitaires St-Luc, Brussels
  - UZ Leuven Gasthuisberg, Leuven
- Bulgaria (2):
  - Shat Np Sveti Naum; 3Rd Clinic of Neurology, Sofia
  - MBAL St. Marina; First Neurology Department, Varna
- Canada (14):
  - University of Calgary; Heritage Medical Research Clinic, Calgary, Alberta
  - True North Clinical Research-Halifax, Halifax, Nova Scotia
  - True North Clinical Research, New Minas, Nova Scotia
  - Jbn Medical Diagnostic Services Inc., Burlington, Ontario
  - Parkwood Hospital; Geriatric Medicine, London, Ontario
  - Kawartha Centre - Redefining Healthy Aging, Peterborough, Ontario
  - Toronto Memory Program, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Recherches Neuro-Hippocame, Gatineau, Quebec
  - NeuroSearch Developpements inc, Greenfield Park, Quebec
  - Jewish General Hospital / McGill University, Montreal, Quebec
  - Centre Hospitalier Affilie Universitaire de Quebec - Hopital de L'Enfant Jesus, Québec, Quebec
  - McGill Univeristy; Douglas Mental Health University Institute; Neurological and Psychiatric, Verdun, Quebec
  - Alpha Recherche Clinique, Québec
- Denmark (2):
  - Aarhus Universitetshospital, Neurologisk Afdeling F, Demensklinikken, Aarhus N
  - Rigshospitalet, Hukommelsesklinikken, Koebenhavn Oe
- Finland (2):
  - University of Eastern Finland, Kuopio
  - CRST Oy, Turku
- France (7):
  - Hopital Pellegrin; Cmrr Aquitaine, Bordeaux
  - Hopital Pierre Wertheimer; Laboratoire De Neuro Psychologie, Bron
  - CHU de Limoges Hopital Dupuytren; Service de Medecine Geriatrique, Limoges
  - CHU de la Timone - Hopital d Adultes; Service de Neurologie, Marseille
  - CHU Rennes - hopital Hotel Dieu; Consultation Memoire - Gerontologie, Rennes
  - Hopital Hautepierre; Centre dInvestigation Clinique, Strasbourg
  - Hopital la Grave; Gerontopole - Centre de Recherche Clinique, Toulouse
- Germany (7):
  - ECRC Experimental and Clinical Research Center, Charité Campus Berlin Buch, Memory Clinic, Berlin
  - PANAKEIA - Arzneimittelforschung Leipzig GmbH, Leipzig
  - Pharmakologisches Studienzentrum, Mittweida
  - Neurologische Praxis Dr. Andrej Pauls, München
  - Klinikum rechts der Isar der TU München; Klinikapotheke, München
  - Universitätsklinikum Ulm; Klinik für Neurologie, Ulm
  - Studienzentrum Nordwest, Dr. med. Joachim Springub / Herr Wolfgang Schwarz, Westerstede
- Semmelweis University; Department of Neurology, Budapest, Hungary
- Italy (7):
  - Nuovo Ospedale Civile S. Agostino-Estense; Clinica Neurologica - Dipartimento di Neuroscienze, Modena, Emilia-Romagna
  - Azienda Ospedaliera Universitaria Policlinico Tor Vergata; Neurologia, Rome, Lazio
  - Umberto I Policlinico di Roma-Università di Roma La Sapienza, Rome, Lazio
  - IRCCS "Centro S. Giovanni di Dio" Fatebenefratelli -UO Alzheimer, Brescia, Lombardy
  - Irccs Multimedica Santa Maria; Unita' Di Neurologia, Castellanza, Lombardy
  - ASST DI MONZA; Neurologia, Monza, Lombardy
  - A.O. Universitaria Pisana; Neurologia, Pisa, Tuscany
- Japan (11):
  - Medical Corporation Hakuyokai Kashiwado Hospital, Chiba
  - National Hospital Organization Chiba-east Hospital; Neurology, Chiba
  - Juntendo University Urayasu Hospital; Neurology, Chiba
  - Fukuoka University Hospital; Neurology and Health Care, Fukuoka
  - Maebashi Red Cross Hospital; Neurology, Gunma
  - National Hospital Organization Hiroshima-Nishi Medical Center, Hiroshima
  - Hyogo Brain and Heart Center at Himeji; Department of Aging Brain and Cognitive Disorders, Hyōgo
  - Shonan Kamakura General Hospital; Neurology, Kanagawa
  - Kurashiki Heisei Hospital; Neurology, Okayama
  - Oita University Hospital; Neurology, Ōita
  - Shizuoka City Shimizu Hospital; Neurology, Shizuoka
- Netherlands (2):
  - Brain Research Center B.V, Amsterdam
  - Erasmus Mc - Locatie Centrum; Dept of Neurology, Rotterdam
- Portugal (2):
  - Hospital Prof. Dr. Fernando Fonseca; Servico de Neurologia, Amadora
  - Hospital de Santa Maria; Servico de Neurologia, Lisbon
- Russia (7):
  - State Autonomous Healthcare Institution "Republican Clinical Neurological Center, Kazan'
  - State autonomous institution of healthcare Inter-regional clinical and diagnostic center, Kazan'
  - Institution of RAMS (Mental Health Research Center of RAMS), Moscow
  - SBEI of HPI The 1st Moscow State Medical University n.a. I.M. Sechenov of MOH of RF, Moscow
  - Saint Petersburg State Institution of Healthcare City Geriatric Medico-Social Center, Saint Petersburg
  - Russian Medical Military Academy n.a. S.M.Kirov; Neurology Department, Saint Petersburg
  - City Clinical Hospital # 2 n.a. V.I. Razumovsky, Saratov
- South Korea (9):
  - Dong-A University Medical Center, Busan
  - Seoul National University Bundang Hospital; Neurology Department, Gyeonggi-do
  - Inha University Hospital; Neurology Department, Incheon
  - Konkuk University Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Ewha Womans University Hospital (Seoul), Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - Asan Medical Center., Seoul
  - Ewha Womans University Mokdong Hospital; Dept of Neurology, Seoul
- Spain (8):
  - Hospital General Universitario de Elche; Servicio de Neurología, Elche, Alicante
  - Fundació ACE, BArcelon, Barcelona
  - Policlínica Guipuzkoa; Servicio de Neurología, Donosti-San Sebastián, Guipuzcoa
  - Hospital de Cruces; Servicio de Neurologia, Barakaldo, Vizcaya
  - Hospital del Mar; Servicio de Neurologia, Barcelona
  - Hospital Universitario 12 de Octubre; Servicio de Neurologia, Madrid
  - Hospital Universitario Virgen Macarena; Servicio de Neurologia, Seville
  - Hospital Universitari i Politecnic La Fe, Valencia
- Sweden (2):
  - Skånes Universitetssjukhus Malmö, Minneskliniken, Malmo
  - KAROLINSKA UNI HOSPITAL, HUDDINGE; Mottagning Kognitiv Forskning, M54, Stockholm
- Switzerland (2):
  - Felix Platter-Spital Medizin Geriatrie, Basel
  - CHUV Lausanne Memory clinique, Lausanne
- Turkey (Türkiye) (3):
  - Istanbul University Istanbul School of Medicine; Neurology, Istanbul
  - Dokuz Eylul University Medicine Faculty; Noroloji Departmani, Izmir
  - Ondokuz Mayis University School of Medicine; Neurology, Samsun
- United Kingdom (6):
  - Sussex Partnership NHS Foundation Trust; Cognitive Treatment and Research unit, Crowborough
  - Glasgow Memory Clinic, Glasgow
  - Charing Cross Hospital; Dept of Neurosciences, London
  - Manchester Royal Infirmary, Manchester
  - Royal Preston Hosptial, Preston
  - Memory Service North, Sheffield

REFERENCES:
- [Derived] Klein G, Delmar P, Voyle N, Rehal S, Hofmann C, Abi-Saab D, Andjelkovic M, Ristic S, Wang G, Bateman R, Kerchner GA, Baudler M, Fontoura P, Doody R. Gantenerumab reduces amyloid-beta plaques in patients with prodromal to moderate Alzheimer's disease: a PET substudy interim analysis. Alzheimers Res Ther. 2019 Dec 12;11(1):101. doi: 10.1186/s13195-019-0559-z. PMID 31831056

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Part 1 of the study was conducted at 116 centers in 21 countries and part 2 was conducted at 75 centers in 17 countries.
Pre-assignment Details: A total of 389 participants were enrolled out of which 387 were randomized and treated (192 received gantenerumab and 195 received placebo) in part 1 of the study. Of these, a total of 230 participants enrolled into Part 2 of the study: 225 participants received at least one dose of study drug. Participants who had discontinued from Part 1 of the study were not allowed to enroll in Part 2.
Groups:
- Part 1: Placebo: Participants received matching placebo by subcutaneous (SC) injection every 4 weeks (Q4W) up to 100 weeks during Part 1 of study.
- Part 1: Gantenerumab: Participants received 105 mg Gantenerumab by SC injection Q4W for 24 weeks and if eligible 225 mg SC injection Q4W from weeks 28-100 during Part 1 of the study.
- Part 2 (OLE Treatment): Placebo Switched to Gantenerumab up to 1200 mg: Participants who had received Placebo in Part 1, received Gantenerumab at doses up to 1200 mg by SC injection Q4W for up to 2 years. Additionally, participants were given the option to continue receiving open-label gantenerumab treatment for 3 years.
Period: Part 1: Double Blind Treatment
Arm/Group | Part 1: Placebo | Part 1: Gantenerumab | Part 2 (OLE Treatment): Placebo Switched to Gantenerumab up to 1200 mg | Part 2 (OLE Treatment): Gantenerumab up to 1200 mg
Started | 195 | 192 | 0 | 0
Completed | 134 | 136 | 0 | 0
Not Completed | 61 | 56 | 0 | 0
Not completed — Death | 3 | 3 | 0 | 0
Not completed — Adverse Event | 2 | 8 | 0 | 0
Not completed — Withdrawal by Subject | 42 | 29 | 0 | 0
Not completed — Physician Decision | 2 | 4 | 0 | 0
Not completed — Lost to Follow-up | 1 | 2 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0
Not completed — Non-Compliance | 2 | 4 | 0 | 0
Not completed — Other | 6 | 3 | 0 | 0
Not completed — Part 1 Terminated by Sponsor | 3 | 2 | 0 | 0
Period: Part 2: Open-label Extension
Arm/Group | Part 1: Placebo | Part 1: Gantenerumab | Part 2 (OLE Treatment): Placebo Switched to Gantenerumab up to 1200 mg | Part 2 (OLE Treatment): Gantenerumab up to 1200 mg
Started | 0 | 0 | 119 | 111
Completed | 0 | 0 | 49 | 50
Not Completed | 0 | 0 | 70 | 61
Not completed — Adverse Event | 0 | 0 | 6 | 8
Not completed — Death | 0 | 0 | 7 | 4
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Non-Compliance | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 39 | 32
Not completed — Study Terminated By Sponsor | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 8 | 5
Not completed — Other | 0 | 0 | 9 | 9

BASELINE CHARACTERISTICS:
Population: The safety-evaluable population consisted of all participants who had received at least one dose of study drug, regardless of whether the participant withdrew prematurely or not.
Groups:
- Part 1: Placebo: Participants received matching placebo by SC injection every 4 weeks Q4W up to 100 weeks during Part 1 of study.
- Total: Total of all reporting groups
Arm/Group | Part 1: Placebo | Part 1: Gantenerumab | Part 2 (OLE Treatment): Placebo Switched to Gantenerumab up to 1200 mg | Part 2 (OLE Treatment): Gantenerumab up to 1200 mg | Total
Number analyzed (Participants) | 195 | 192 | 117 | 108 | 612
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Part 1 of the study.
  years
    number analyzed (Participants) | 195 | 192 | 0 | 0 | 387
    (all) | 70.1 (8.6) | 69.7 (8.9) |  |  | 69.9 (8.7)
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Part 2 of the study.
  years
    number analyzed (Participants) | 0 | 0 | 117 | 108 | 225
    (all) |  |  | 71.82 (8.09) | 71.01 (9.31) | 71.43 (8.69)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Part 1 of the study.
  Participants
    number analyzed (Participants) | 195 | 192 | 0 | 0 | 387
    Female | 113 | 98 |  |  | 211
    Male | 82 | 94 |  |  | 176
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Part 2 of the study.
  Participants
    number analyzed (Participants) | 0 | 0 | 117 | 108 | 225
    Female |  |  | 69 | 61 | 130
    Male |  |  | 48 | 47 | 95
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Part 1 of the study.
  Participants
    number analyzed (Participants) | 195 | 192 | 0 | 0 | 387
    Hispanic or Latino | 11 | 12 |  |  | 23
    Not Hispanic or Latino | 178 | 176 |  |  | 354
    Unknown or Not Reported | 6 | 4 |  |  | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Part 2 of the study.
  Participants
    number analyzed (Participants) | 0 | 0 | 117 | 108 | 225
    Hispanic or Latino |  |  | 9 | 10 | 19
    Not Hispanic or Latino |  |  | 108 | 96 | 204
    Unknown or Not Reported |  |  | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Part 1 of the study.
  Participants
    number analyzed (Participants) | 195 | 192 | 0 | 0 | 387
    American Indian or Alaska Native | 0 | 0 |  |  | 0
    Asian | 23 | 21 |  |  | 44
    Native Hawaiian or Other Pacific Islander | 0 | 1 |  |  | 1
    Black or African American | 2 | 2 |  |  | 4
    White | 164 | 166 |  |  | 330
    More than one race | 1 | 0 |  |  | 1
    Unknown or Not Reported | 5 | 2 |  |  | 7
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Part 2 of the study.
  Participants
    number analyzed (Participants) | 0 | 0 | 117 | 108 | 225
    American Indian or Alaska Native |  |  | 0 | 0 | 0
    Asian |  |  | 19 | 19 | 38
    Native Hawaiian or Other Pacific Islander |  |  | 0 | 1 | 1
    Black or African American |  |  | 2 | 2 | 4
    White |  |  | 94 | 85 | 179
    More than one race |  |  | 0 | 0 | 0
    Unknown or Not Reported |  |  | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Part 2: Percentage of Participants With Adverse Events (AEs) or Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. SAE is any adverse event that is fatal or which requires or prolongs inpatient hospitalization or results in persistent or significant disability/incapacity or causes congenital anomaly/birth defect or results in a significant medical event in the investigator's judgment.
Time Frame: First dose up to 4 weeks after the last dose of study drug (up to 249 weeks)
Population: as for baseline characteristics
Measure: Number; unit: Percentage of Participants
Arm/Group | Part 2 (OLE Treatment): Placebo Switched to Gantenerumab up to 1200 mg | Part 2 (OLE Treatment): Gantenerumab up to 1200 mg
Number analyzed (Participants) | 117 | 108
Percentage of Participants
  AEs | 91.5 | 95.4
  SAEs | 24.8 | 38.0

2. Primary Outcome: Part 2: Percentage of Participants With Treatment Emergent Anti-Drug Antibodies (ADAs)
Description: Participants were considered positive or negative for ADA based on their baseline and post-baseline sample results. The number and percentage of participants with confirmed positive ADA levels were determined for participants previously (in part 1) on Gantenerumab and Placebo. The prevalence of ADA at baseline was calculated as the percentage of participants with confirmed positive ADA levels at baseline relative to the total number of participants with a sample available at baseline. The incidence of treatment-emergent ADAs was determined as the percentage of participants with confirmed post-baseline positive ADAs relative to the total number of participants that had at least one post-baseline sample available for ADA analysis.
Time Frame: First dose up to last dose (Baseline up to until maximum 5 years)
Population: The safety population consisted of all participants who had received at least one dose of study drug, regardless of whether the participants withdrew prematurely or not. The number of participants analyzed indicates the number of participants evaluated for the outcome measure.
Measure: Number; unit: Percentage of Participants
Arm/Group | Part 2 (OLE Treatment): Placebo Switched to Gantenerumab up to 1200 mg | Part 2 (OLE Treatment): Gantenerumab up to 1200 mg
Number analyzed (Participants) | 115 | 106
Percentage of Participants | 2.6 | 2.8

3. Primary Outcome: Part 2: Percentage of Participants With Adverse Events Leading to Discontinuation of Treatment
Description: Percentage of participants with adverse events leading to discontinuation from treatment were reported.
Time Frame: First dose up to 4 weeks after the last dose in OLE (Up to approximately 249 weeks)
Population: The safety population consisted of all participants who had received at least one dose of study drug, regardless of whether the participants withdrew prematurely or not.
Measure: Number; unit: Percentage of Participants
Arm/Group | Part 2 (OLE Treatment): Placebo Switched to Gantenerumab up to 1200 mg | Part 2 (OLE Treatment): Gantenerumab up to 1200 mg
Number analyzed (Participants) | 117 | 108
Percentage of Participants | 12.0 | 15.7

4. Secondary Outcome: Part 1: Percentage of Participants With AEs, SAEs
Description: An AE is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. A serious adverse event is any adverse event that is fatal or which requires or prolongs inpatient hospitalization or results in persistent or significant disability/incapacity or causes congenital anomaly/birth defect or results in a significant medical event in the investigator's judgment.
Time Frame: First dose up to last dose (Up to approximately 152 weeks)
Population: The safety population consisted of all participants who received at least one dose of study drug, regardless of whether the participants withdrew prematurely or not.
Measure: Number; unit: Percentage of Participants
Arm/Group | Part 1: Placebo | Part 1: Gantenerumab
Number analyzed (Participants) | 195 | 192
Percentage of Participants
  AEs | 80.5 | 82.8
  SAEs | 12.3 | 12.0

5. Secondary Outcome: Part 1: Percentage of Participants With Treatment Emergent ADAs
Description: as for outcome 2
Time Frame: First dose up to last dose (Up to approximately 152 weeks)
Population: The safety population consisted of all participants who received at least one dose of study drug, regardless of whether the participants withdrew prematurely or not. The number of participants analyzed indicates the number of participants evaluated for the outcome measure.
Measure: Number; unit: Percentage of Participants
Arm/Group | Part 1: Placebo | Part 1: Gantenerumab
Number analyzed (Participants) | 194 | 191
Percentage of Participants | 3.6 | 11.5

6. Secondary Outcome: Part 1: Gantenerumab Plasma Concentration at Multiple Timepoints
Time Frame: Pre-dose: Weeks 4, 8, 12, 24, 48, 72 and Post dose: Day 4
Population: The pharmacokinetic (PK) evaluable population consisted of all participants that were treated with gantenerumab and provided at least 1 post-baseline PK sample. Number analyzed is the number of participants with data available for analyses at the given time-point.
Measure: Mean (Standard Deviation); unit: μg/mL
Groups:
- Gantenerumab: Participants received 105 mg Gantenerumab by SC injection Q4W for 24 weeks and if eligible 225 mg SC injection Q4W from weeks 28-100 during Part 1 of the study.
Arm/Group | Gantenerumab
Number analyzed (Participants) | 192
μg/mL
  Day 4: number analyzed (Participants) | 183
  Day 4 | 4.11 (2.59)
  Week 4: number analyzed (Participants) | 190
  Week 4 | 2.06 (0.89)
  Week 8: number analyzed (Participants) | 188
  Week 8 | 3.11 (1.41)
  Week 12: number analyzed (Participants) | 184
  Week 12 | 3.35 (1.63)
  Week 24: number analyzed (Participants) | 177
  Week 24 | 3.71 (2.13)
  Week 48: number analyzed (Participants) | 137
  Week 48 | 7.61 (3.88)
  Week 72: number analyzed (Participants) | 79
  Week 72 | 7.66 (4.44)

7. Secondary Outcome: Part 1: Percentage of Participants With Adverse Events Leading to Discontinuation of Treatment
Description: Percentage of participants with adverse events leading to discontinuation from treatment were reported.
Time Frame: First dose up to last dose (Up to approximately 152 weeks)
Population: as for outcome 4
Measure: Number; unit: Percentage of Participants
Arm/Group | Part 1: Placebo | Part 1: Gantenerumab
Number analyzed (Participants) | 195 | 192
Percentage of Participants | 2.6 | 6.8

8. Secondary Outcome: Part 2: Percent Change From Baseline in Hippocampal Volume at Week 104
Description: Change from baseline in hippocampal right volume (HRV) and hippocampal left volume (HLV) were analyzed at Week 104 using magnetic resonance imaging.
Time Frame: Baseline (Part 1 screening), Week 104
Population: The safety population consisted of all participants who received at least one dose of gantenerumab during the OLE and also had at least one post baseline MRI. The number of participants analyzed indicates the number of participants evaluated for the outcome measure. Number analyzed is the number of participants with data available for analyses at the given time-point.
Measure: Mean (Standard Deviation); unit: Percent Change
Groups:
- Part 2 (OLE Treatment): Gantenerumab up to 1200 mg: Participants who had received Gantenerumab by SC injection in Part 1, received treatment at doses up to 1200 mg by SC injection Q4W for up to 2 years. Additionally, participants were given the option to continue receiving open-label gantenerumab treatment for 3 years.
Arm/Group | Part 2 (OLE Treatment): Placebo Switched to Gantenerumab up to 1200 mg | Part 2 (OLE Treatment): Gantenerumab up to 1200 mg
Number analyzed (Participants) | 52 | 44
Percent Change
  Hippocampal Left Volume- Percent Change at Week 104: number analyzed (Participants) | 50 | 43
  Hippocampal Left Volume- Percent Change at Week 104 | -11.24 (4.04) | -12.10 (4.45)
  Hippocampal Right Volume- Percent Change at Week 104 | -12.49 (4.03) | -11.34 (4.41)

9. Secondary Outcome: Part 2: Percent Change From Baseline in Whole Brain Volume at Week 104
Description: Change from baseline brain volume were analyzed at Week 104 using magnetic resonance imaging.
Time Frame: Baseline (Part 1 screening), Week 104
Population: The safety population consisted of all participants who received at least one dose of gantenerumab during the OLE and also had at least one post baseline MRI. The number of participants analyzed indicates the number of participants evaluated for the outcome measure.
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Part 2 (OLE Treatment): Placebo Switched to Gantenerumab up to 1200 mg | Part 2 (OLE Treatment): Gantenerumab up to 1200 mg
Number analyzed (Participants) | 54 | 44
Percent Change | -4.89 (1.90) | -4.91 (1.58)

10. Secondary Outcome: Part 2: Percent Change From Baseline in Cortical Thickness at Week 104
Description: Change from baseline in cortical thickness were analyzed at Week 104 using magnetic resonance imaging.
Time Frame: Baseline (Part 1 screening), Week 104
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Part 2 (OLE Treatment): Placebo Switched to Gantenerumab up to 1200 mg | Part 2 (OLE Treatment): Gantenerumab up to 1200 mg
Number analyzed (Participants) | 54 | 44
Percent Change | -5.84 (2.33) | -5.58 (1.87)

11. Secondary Outcome: Part 2: Ventricular Volume as Measured by MRI at Week 104
Description: Ventricular volume were analyzed at Week 104 using magnetic resonance imaging.
Time Frame: Part 2: Week 104
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Part 2 (OLE Treatment): Placebo Switched to Gantenerumab up to 1200 mg | Part 2 (OLE Treatment): Gantenerumab up to 1200 mg
Number analyzed (Participants) | 63 | 52
mL | 86.70 (38.37) | 86.21 (30.49)

12. Secondary Outcome: Part 2: Gantenerumab Plasma Concentration at Multiple Timepoints
Time Frame: Pre-dose: Weeks 104, 116, 156, 208; Post-dose: Weeks 53, 101
Population: Of the 225 participants in the OLE safety evaluable population, evaluable PK information was available from 223 participants. The PK evaluable population consisted of all participants that were treated with gantenerumab and provided at least 1 post-baseline PK sample. Number analysed is the number of participants with data available for analyses at the given time-point.
Measure: Mean (Standard Deviation); unit: μg/mL
Groups:
- Part 2 (OLE Treatment): Gantenerumab 1200 mg: Participants who had received placebo or gantenerumab in Part 1, received gantenerumab at doses up to 1200 mg by SC injection Q4W for up to 2 years. Additionally, participants were given the option to continue receiving open-label gantenerumab treatment for 3 years.
Arm/Group | Part 2 (OLE Treatment): Gantenerumab 1200 mg
Number analyzed (Participants) | 223
μg/mL
  Week 53: number analyzed (Participants) | 128
  Week 53 | 80.6 (38.4)
  Week 101: number analyzed (Participants) | 111
  Week 101 | 89.1 (33.6)
  Week 104: number analyzed (Participants) | 141
  Week 104 | 43.5 (22.4)
  Week 116: number analyzed (Participants) | 15
  Week 116 | 3.66 (2.29)
  Week 156: number analyzed (Participants) | 80
  Week 156 | 45.2 (22.5)
  Week 208: number analyzed (Participants) | 48
  Week 208 | 55.8 (37.9)

13. Secondary Outcome: Part 2: Change From Baseline in Brain Amyloid Load at Week 156 in a Subset of Participants
Description: Brain amyloid load over time was assessed using a Florbetapir [F18] injection, a positron emission tomography (PET) radioligand selective to amyloid. Analysis was conducted in a subset of participants who signed consent to participate in the PET substudy. Amyloid PET burden was measured in a composite region of interest (ROI) by using standardized uptake value ratio (SUVR) mapped to the centiloid scale. The composite region was composed of the following six bilateral regions: frontal lobe, parietal lobe, temporal lobe, posterior cingulate cortex, anterior cingulate cortex. The reference region used to normalize the composite region was the cerebellar cortex. SUVR is ratio of tracer uptake in each of cingulate, frontal, parietal and temporal cortexes relative to cerebellum. The centiloid scale anchor points are 0 and 100, where 0 represents a high-certainty amyloid negative scan and 100 represents the amount of global amyloid deposition found in a typical AD scans.
Time Frame: Baseline, Week 156
Population: The safety population consisted of all participants who had received at least one dose of study drug, regardless of whether the participants withdrew prematurely or not. The number of participants analysed indicates the number of participants evaluated for the outcome measure.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Part 2 (OLE Treatment): Placebo Switched to Gantenerumab up to 1200 mg | Part 2 (OLE Treatment): Gantenerumab up to 1200 mg
Number analyzed (Participants) | 13 | 8
Score on a scale | -81.01 (47.08) | -84.93 (28.38)

14. Other Pre Specified Outcome: Part 1: Mean Change From Baseline in Alzheimer's Disease Activity Scale-Cognitive Subscale 13 (ADAS-Cog13) Scores at Week 104
Time Frame: Baseline, Week 104
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Part 1: Mean Change From Baseline in Alzheimer's Disease Cooperative Study-Activities of Daily Living (ADCS-ADL) Scores at Week 104
Time Frame: Baseline, Week 104
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Part 1: Percentage Change From Baseline in Total Tau (T-tau) in CSF at Week 104
Time Frame: Baseline, Week 104
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Part 1: Percentage Change From Baseline in Abeta 1-42 Levels in CSF at Week 104
Time Frame: Baseline, Week 104
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Part 1: Percentage Change From Baseline in Phosphorylated Tau [P-tau] in CSF at Week 104
Time Frame: Baseline, Week 104
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Part 1: Percent Change From Baseline in Hippocampal Volume at Week 104
Time Frame: Baseline, Week 104
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Part 1: Percent Change From Baseline in Whole Brain Volume at Week 104
Time Frame: Baseline, Week 104
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Part 1: Percent Change From Baseline in Cortical Thickness at Week 104
Time Frame: Baseline, Week 104
Reporting Status: Not Posted

22. Other Pre Specified Outcome: Part 1: Ventricular Volume as Measured by MRI at Week 104
Time Frame: Baseline, Week 104
Reporting Status: Not Posted

23. Other Pre Specified Outcome: Part 1: Change From Baseline in Clinical Dementia Rating Global Score (CDR-GS) at Week 104
Time Frame: Baseline, Week 104
Reporting Status: Not Posted

24. Other Pre Specified Outcome: Part 1: Change From Baseline in CDR Sum of Boxes (SB) at Week 104
Time Frame: Baseline, Week 104
Reporting Status: Not Posted

25. Other Pre Specified Outcome: Part 1: Change From Baseline in Neuropsychiatric Inventory (NPI) Total Score at Week 104
Time Frame: Baseline, Week 104
Reporting Status: Not Posted

26. Other Pre Specified Outcome: Part 1: Change From Baseline in NPI Domain Score at Week 104
Time Frame: Baseline, Week 104
Reporting Status: Not Posted

27. Other Pre Specified Outcome: Part 1: Change From Baseline in Mini Mental State Examination (MMSE) Total Score at Week 104
Time Frame: Baseline, Week 104
Reporting Status: Not Posted

28. Other Pre Specified Outcome: Part 1: Change From Baseline in Alzheimer's Dementia (QoL-AD) Global Score at Week 104
Time Frame: Baseline, Week 104
Reporting Status: Not Posted

29. Other Pre Specified Outcome: Part 1: Change From Baseline in Symptom Guide Facilitated (GAS) at Week 104
Time Frame: Baseline, Week 104
Reporting Status: Not Posted

30. Other Pre Specified Outcome: Part 1: Change From Baseline in Dependence Scale (DS) at Week 104
Time Frame: Baseline, Week 104
Reporting Status: Not Posted

31. Other Pre Specified Outcome: Part 1: Change From Baseline in Resource Utilization Dementia-Lite (RUD - Lite) Scale at Week 104
Time Frame: Baseline, Week 104
Reporting Status: Not Posted

32. Other Pre Specified Outcome: Part 1: Change From Baseline in Zarit Caregiver Interview for Alzheimer's Disease (ZCI-AD) at Week 104
Time Frame: Baseline, Week 104
Reporting Status: Not Posted

33. Other Pre Specified Outcome: Part 1: Time to Clinical Decline
Time Frame: Baseline up to Week 104
Reporting Status: Not Posted

34. Other Pre Specified Outcome: Part 1: Change From Baseline in Clinical Composite Score (Prespecified Items From The ADAS-Cog, MMSE, and CDR) at Week 104
Time Frame: Baseline, Week 104
Reporting Status: Not Posted

35. Other Pre Specified Outcome: Part 1: Percentage of Participants With ADAS-Cog Response
Time Frame: Baseline up to Week 152
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Baseline up to 52 weeks after the last dose of study drug (up to 7 years)
Description: The safety-evaluable population consisted of all participants who had received at least one dose of study drug, regardless of whether the participant withdrew prematurely or not.
Arm/Group | Part 1: Placebo | Part 1: Gantenerumab | Part 2 (OLE Treatment): Placebo Switched to Gantenerumab up to 1200 mg | Part 2 (OLE Treatment): Gantenerumab up to 1200 mg
All-Cause Mortality (participants affected / at risk) | 11/195 | 8/192 | 5/117 | 5/108
Serious Adverse Events (participants affected / at risk) | 53/195 | 61/192 | 29/117 | 41/108
Other Adverse Events (participants affected / at risk) | 147/195 | 159/192 | 94/117 | 91/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Placebo (N=195) | Part 1: Gantenerumab (N=192) | Part 2 (OLE Treatment): Placebo Switched to Gantenerumab up to 1200 mg (N=117) | Part 2 (OLE Treatment): Gantenerumab up to 1200 mg (N=108)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 3 (3) | 0 (0) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Ocular hypertension (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cyst (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Anaphylactic shock (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Appendiceal abscess (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Bacterial sepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Colonic abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis rotavirus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Periodontitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 1 (1) | 2 (2) | 1 (1)
Respiratory tract infection (Infections and infestations) | 3 (3) | 0 (0) | 3 (3) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Shunt infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tonsillitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3) | 3 (3) | 3 (3) | 2 (2)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (2) | 1 (1) | 0 (0) | 1 (1)
Chest injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Comminuted fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 5 (5) | 0 (0) | 3 (3)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Jaw fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Multiple fractures (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Optic nerve injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Subdural haematoma (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 1 (1) | 2 (2)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram abnormal (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Cerebellar tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Ovarian epithelial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of pharynx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ARIA-E (Nervous system disorders) | 2 (2) | 2 (3) | 2 (2) | 2 (2)
ARIA-H (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Brain stem infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cerebral haematoma (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cerebral venous sinus thrombosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dementia Alzheimer's type (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Dementia of the Alzheimer's type, with delusions (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hemiplegia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Leukoencephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nervous system disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neurotoxicity (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Psychomotor hyperactivity (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 2 (2) | 1 (1) | 2 (2)
Transient ischaemic attack (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Vertebral artery dissection (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vertebrobasilar stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Affective disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aggression (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 1 (2) | 0 (0) | 1 (2)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Psychotic symptom (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Suicide threat (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aortic aneurysm rupture (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Giant cell arteritis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Placebo (N=195) | Part 1: Gantenerumab (N=192) | Part 2 (OLE Treatment): Placebo Switched to Gantenerumab up to 1200 mg (N=117) | Part 2 (OLE Treatment): Gantenerumab up to 1200 mg (N=108)
Constipation (Gastrointestinal disorders) | 14 (15) | 16 (20) | 6 (7) | 12 (15)
Diarrhoea (Gastrointestinal disorders) | 23 (27) | 11 (18) | 11 (14) | 8 (13)
Nausea (Gastrointestinal disorders) | 15 (24) | 10 (11) | 3 (9) | 4 (4)
Vomiting (Gastrointestinal disorders) | 11 (16) | 14 (18) | 6 (11) | 6 (7)
Injection site reaction (General disorders) | 49 (284) | 52 (322) | 48 (281) | 44 (280)
Oedema peripheral (General disorders) | 2 (2) | 10 (11) | 1 (1) | 8 (9)
Pyrexia (General disorders) | 4 (4) | 7 (9) | 2 (2) | 6 (8)
Bronchitis (Infections and infestations) | 10 (13) | 10 (11) | 6 (9) | 5 (6)
Influenza (Infections and infestations) | 8 (10) | 14 (19) | 4 (4) | 10 (12)
Nasopharyngitis (Infections and infestations) | 27 (35) | 23 (31) | 13 (14) | 11 (15)
Upper respiratory tract infection (Infections and infestations) | 20 (30) | 7 (12) | 10 (13) | 3 (5)
Urinary tract infection (Infections and infestations) | 17 (20) | 18 (28) | 11 (13) | 7 (14)
Contusion (Injury, poisoning and procedural complications) | 12 (15) | 16 (21) | 5 (7) | 8 (9)
Fall (Injury, poisoning and procedural complications) | 28 (44) | 35 (69) | 16 (25) | 22 (41)
Skin abrasion (Injury, poisoning and procedural complications) | 6 (7) | 12 (17) | 3 (3) | 5 (10)
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 (15) | 13 (23) | 8 (8) | 7 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 20 (21) | 17 (19) | 8 (9) | 5 (5)
Neck pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 2 (2) | 6 (6) | 1 (1)
ARIA-E (Nervous system disorders) | 32 (42) | 42 (70) | 29 (35) | 30 (51)
ARIA-H (Nervous system disorders) | 30 (39) | 36 (42) | 19 (23) | 23 (27)
Dizziness (Nervous system disorders) | 18 (24) | 17 (26) | 13 (13) | 6 (6)
Headache (Nervous system disorders) | 29 (38) | 22 (44) | 15 (18) | 12 (24)
Agitation (Psychiatric disorders) | 13 (16) | 18 (21) | 9 (10) | 8 (9)
Anxiety (Psychiatric disorders) | 13 (13) | 13 (14) | 5 (5) | 6 (6)
Depression (Psychiatric disorders) | 17 (17) | 13 (14) | 8 (8) | 2 (2)
Insomnia (Psychiatric disorders) | 12 (15) | 15 (16) | 7 (8) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 9 (9) | 12 (12) | 4 (4) | 5 (5)
Hypertension (Vascular disorders) | 13 (13) | 13 (15) | 4 (4) | 5 (5)

LIMITATIONS AND CAVEATS:
As the participants transitioned early to OLE, most participants did not reach the primary analysis timepoint (Week 104). Hence, the efficacy endpoints for Part 1 became exploratory in nature.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2020-02-28): https://cdn.clinicaltrials.gov/large-docs/08/NCT02051608/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-31): https://cdn.clinicaltrials.gov/large-docs/08/NCT02051608/SAP_001.pdf